CLINICAL TRIAL: NCT05107986
Title: Outcomes of Laparoscopic Repair in Complicated Groin Hernia: a Single Institutional Based Cohort Study in Nepal
Brief Title: Laparoscopy in Complicated Groin Hernia
Status: Completed | Type: Observational
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Bhawani Khanal, Asisstant Professor, B.P. Koirala Institute of Health Sciences
Other Study IDs: IRC/1217/018
Record Dates: First submitted 2021-10-07; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Inguinal Hernia
Keywords: Complicated groin hernia; Totally extra-peritoneal repair; Transabdominal preperitoneal repair
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with complicated groin hernia
  Interventions: Procedure: laparoscopic repair

INTERVENTIONS:
Procedure: laparoscopic repair — All patients of cohort underwent laparoscopic repair.

SUMMARY:
This study assessed the outcomes of laparoscopic repair in complicated groin hernia. Laparoscopic approach in cases of complicated groin hernia can achieve desirable patient outcomes without major complications, provided good patient selection and expertise. This study provides an insight to the outcomes from the procedure in low resource setting of Nepal.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age greater than 18 years with diagnosis of complicated groin hernia

Exclusion Criteria:

* Patients with features of peritonitis, history of previous abdominal surgery and those unfit for general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of complicated groin hernia
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
intraoperative complications | during surgical procedure
  1. Bleeding (epigastric / testicular vessels) 2. Bowel injury 3. Peritoneal tear
Postoperative complications | upto 6 months post operatively
  1. Seroma 2.Urinary Retention 3. Wound infection

CONTACTS AND LOCATIONS:
Locations (1):
- BP Koirala Institute of Health Sciences, Dharān, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: No